CLINICAL TRIAL: NCT04908605
Title: Emergence Agitation After Nasal Surgery: a Randomized Controlled Comparison Between Melatonin and Mirtazapine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS251 /202l
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Mirtazapine; Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirtazapine group (Group I) (n=55) (Active Comparator)
  Interventions: Drug: Mirtazapine
- Melatonin group (Group II) (n=55) (Active Comparator)
  Interventions: Drug: Melatonin
- Placebo group (Group III) (n=55) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — Every patient will be given mirtazapine 30 mg tablet
  Arms: Mirtazapine group (Group I) (n=55)
Drug: Melatonin — Every patient will be given melatonin 5 mg tablet
  Arms: Melatonin group (Group II) (n=55)
Drug: Placebo — Every patient will be given a matching placebo tablet
  Arms: Placebo group (Group III) (n=55)

SUMMARY:
Emergence agitation (EA) is common after nasal surgery under general anesthesia, which can lead to several problems, such as increased risk of injury to the patient or medical staff, pain, decreased patient satisfaction, hemorrhage, re-bleeding at the operation site and unplanned self-extubation.

Melatonin is an oral or sublingual medication, most commonly used for insomnia and improving sleep in different conditions for example shift-work disorder and for helping people to establish a day and night cycle especially blind children or adults.

Mirtazapine is an antidepressant used in medicine in a pill form, most commonly used for major depressive disorder and other mood disorders, relief of anxiety, panic disorders, insomnia, headache and migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients according to American Society of Anesthesiologists physical status classification (ASA) I or II.
2. Patients according to Mallampati classification I or II.
3. Patients accepting the study and consenting.
4. Undergoing general anesthesia for elective nasal surgery in which nasal packing on each side was used until 24 h after surgery.
5. Body mass index(BMI)<30

Exclusion Criteria:

1. Patient's refusal.
2. Known allergy to any of the study medications.
3. History of obstructive sleep apnea.
4. History of psychiatric illness or intake of antipsychotics.
5. History of liver impairment.
6. Pregnancy.
7. History of uncontrolled hypertension.
8. History of renal disease.
9. Body mass index (BMI) ≥30 kg/m2.
10. Contraceptive drugs.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Total number of patients with the Riker sedation-agitation score ≥5 | 24 hours postoperatively
  Total number of patients with the Riker sedation-agitation score ≥5

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No